CLINICAL TRIAL: NCT04870411
Title: Immunological Response to COVID-19 Vaccine in Patients With Autoimmune and Inflammatory Diseases Treated With Immunosuppressants and/or Biologics
Acronym: COVADIS
Status: Terminated | Type: Observational
Why Stopped: Most of the patients were already vaccinated
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Immunov (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210167; 2021-A00181-40 (Other: France : ANSM)
Record Dates: First submitted 2021-03-26; First posted 2021-05-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Diseases; Inflammatory Disorder
Keywords: Covid-19; vaccine; SARS-CoV2; autoimmune diseases; immunosuppressants
MeSH Terms: conditions — Autoimmune Diseases; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with auto-immune or autoinflammatory diseases: Patients with auto-immune or autoinflammatory diseases treated with immunosuppressants and/or biologics
  Interventions: Biological: Blood sample
- Patients without auto-immune or autoinflammatory diseases: Patients without auto-immune or autoinflammatory diseases and not treated with immunosuppressants and/or biologics
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Humoral and cellular immune response. Sample before vaccination, 1 month, 3 months, 6 months and 12 months post-vaccination

SUMMARY:
Vaccination against the new coronavirus (SARS-CoV-2) was extended to patients at risk of severe forms of Covid-19, including in particular patients with autoimmune and inflammatory diseases treated by immunosuppressants and/or biologics.

In this particular population, the effectiveness of vaccines, in particular influenza and pneumococcal vaccinations, is often reduced, especially in case of treatment with rituximab and / or methotrexate.

Regarding the SARS-CoV-2 vaccine, the studies that allowed the marketing authorization of the available vaccines did not include patients treated with immunosuppressants or immunomodulators.

Thus, the impact of treatments on the production of neutralizing antibodies and specific T lymphocytes is not known.

The goal of this study is to assess the immune response to the SARS-CoV-2 vaccine in patients with autoimmune and inflammatory diseases treated with immunosuppressants or immunomodulators.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 :
* Patient over 18 years old,
* Patient informed and not opposed to participate
* Patient followed for an autoimmune or inflammatory disease (vasculitis, systemic lupus, systemic sclerosis, non-infectious uveitis)
* Treatment with immunosuppressant and / or immunomodulator
* Group 2 :
* Patient over 18 years old,
* Patient informed and not opposed to participate
* Patient not followed for an autoimmune or inflammatory disease (vasculitis, systemic lupus, systemic sclerosis, non-infectious uveitis)
* Absence of treatment with immunosuppressant and / or immunomodulator

Exclusion Criteria:

* Contraindication to vaccination
* Progressive cancer
* Pregnant or breastfeeding woman
* Current infection less than 3 weeks old
* Weight less than 40 kg
* Patient under tutor- or curator-ship
* Patient without health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with auto-immune or autoinflammatory diseases treated with immunosuppressants and/or biologics = 170 patients Patients without auto-immune or autoinflammatory diseases and not treated with immunosuppressants and/or biologics = 30 patients
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with neutralizing antibody | 1 month after vaccination

SECONDARY OUTCOMES:
Proportion of patients with neutralizing antibody | 3 months after vaccination
Proportion of patients with neutralizing antibody | 6 months after vaccination
Proportion of patients with neutralizing antibody | 12 months after vaccination
Proportion of patients with anti-SARS-CoV2 specific T lymphocytes | 1 month after vaccination
Proportion of patients with anti-SARS-CoV2 specific T lymphocytes | 3 months after vaccination
Proportion of patients with anti-SARS-CoV2 specific T lymphocytes | 6 months after vaccination
Proportion of patients with anti-SARS-CoV2 specific T lymphocytes | 12 months after vaccination
Proportion of patients with symptomatic infection by Covid 19 during follow-up | 1 month after vaccination
Proportion of patients with symptomatic infection by Covid 19 during follow-up | 3 months after vaccination
Proportion of patients with symptomatic infection by Covid 19 during follow-up | 6 months after vaccination
Proportion of patients with symptomatic infection by Covid 19 during follow-up | 12 months after vaccination
Proportion of patients with neutralizing antibody and anti-SARS-CoV2 specific T cells according to the immunosuppressive or immunomodulative treatment | 1 month after vaccination
Proportion of patients with neutralizing antibody and anti-SARS-CoV2 specific T cells according to the immunosuppressive or immunomodulative treatment | 3 months after vaccination
Proportion of patients with neutralizing antibody and anti-SARS-CoV2 specific T cells according to the immunosuppressive or immunomodulative treatment | 6 months after vaccination
Proportion of patients with neutralizing antibody and anti-SARS-CoV2 specific T cells according to the immunosuppressive or immunomodulative treatment | 12 months after vaccination
Proportion of patients with flair of autoimmune disease | 1 month after vaccination
Proportion of patients with flair of autoimmune disease | 3 months after vaccination
Proportion of patients with flair of autoimmune disease | 6 months after vaccination
Proportion of patients with flair of autoimmune disease | 12 months after vaccination
Proportion of patients with treatment-related adverse events grade 3 or 4 | 1 month after vaccination
Proportion of patients with treatment-related adverse events grade 3 or 4 | 3 months after vaccination
Proportion of patients with treatment-related adverse events grade 3 or 4 | 6 months after vaccination
Proportion of patients with treatment-related adverse events grade 3 or 4 | 12 months after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Internal medicine Service - Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Welzel D, Roskamm N, Samek L, Sturzenhofecker P. Pindolol postmyocardial infarction study: evaluation of the drug's antiarrhythmic and antianginal activity. Am Heart J. 1982 Aug;104(2 Pt 2):512-5. doi: 10.1016/0002-8703(82)90148-x. PMID 7102538
- [Background] Cameron MM, Milligan PJ, Llanos-Cuentas A, Davies CR. An association between phlebotomine sandflies and aphids in the Peruvian Andes. Med Vet Entomol. 1995 Apr;9(2):127-32. doi: 10.1111/j.1365-2915.1995.tb00168.x. PMID 7787219
- [Background] Scholes J, Freeman M. The reflective dialogue and repertory grid: a research approach to identify the unique contribution of nursing, midwifery or health visiting to the therapeutic milieu. J Adv Nurs. 1994 Nov;20(5):885-93. doi: 10.1046/j.1365-2648.1994.20050885.x. PMID 7745181
- [Background] Sacre K, Goulenok T, Bahuaud M, Francois C, Van der Haegen MC, Alexandra JF, Aucouturier P, Hurtado-Nedelec M, Moins-Teisserenc H, Batteux F, Papo T. Impaired long-term immune protection following pneumococcal 13-valent/23-valent polysaccharide vaccine in systemic lupus erythematosus (SLE). Ann Rheum Dis. 2018 Oct;77(10):1540-1542. doi: 10.1136/annrheumdis-2017-212789. Epub 2018 Feb 14. No abstract available. PMID 29444908
- [Background] Hadjadj J, Planas D, Ouedrani A, Buffier S, Delage L, Nguyen Y, Bruel T, Stolzenberg MC, Staropoli I, Ermak N, Macraigne L, Morbieu C, Henriquez S, Veyer D, Pere H, Casadevall M, Mouthon L, Rieux-Laucat F, Chatenoud L, Schwartz O, Terrier B. Immunogenicity of BNT162b2 vaccine against the Alpha and Delta variants in immunocompromised patients with systemic inflammatory diseases. Ann Rheum Dis. 2022 May;81(5):720-728. doi: 10.1136/annrheumdis-2021-221508. Epub 2022 Jan 12. PMID 35022159